CLINICAL TRIAL: NCT01876940
Title: A Randomized Comparison of Free-handed Fiberoptic Intubation Compared With Fiberoptic Intubation Through an Air-QTM Intubating Laryngeal Airway in Children Less Than Two Years of Age: Does Operator Experience Affect Time to Successful Tracheal Intubation?
Brief Title: Comparison of Fiberoptic Intubation With Fiberoptic Intubation Through an Air-Q Intubating Laryngeal Airway in Infants and Small Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB#2013-15391
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Fiberoptic Intubation in Children
Keywords: supraglottic airway; children; tracheal intubation; fiberoptic bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fiberoptic Intubation performed by an expert (Active Comparator): Tracheal intubation will be performed by an expert anesthesia attending with and without use of the air-Q
  Interventions: Device: air-Q, followed by fiberoptic intubation; Device: Free-hand Fiberoptic Intubation
- Fiberoptic Intubation performed by a novice (Experimental): Tracheal intubation will be performed by an anesthesia trainee with and without use of the air-Q
  Interventions: Device: air-Q, followed by fiberoptic intubation; Device: Free-hand Fiberoptic Intubation

INTERVENTIONS:
Device: air-Q, followed by fiberoptic intubation
  Other Names: Device will be placed and fiberoptic tracheal intubation will be performed and timed. Laryngeal grade of view will also be assessed
Device: Free-hand Fiberoptic Intubation — Fiberoptic tracheal intubation will be performed without use of the air-Q and timed. Laryngeal grade of view will also be assessed

SUMMARY:
The goal of this prospective randomized study is to compare the effect of operator experience on the ability to use fiberoptic-guided intubation in children less than two years old, with and without the use of an air-Q as a conduit. The question the investigators are trying to answer is: Does the operator experience make a significant difference in the time for successful fiberoptic guided tracheal intubation with and without the use of an air-Q intubating laryngeal airway?

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of operator experience on the ability to use fiberoptic-guided intubation in children less than two years old, with and without the use of an air-Q as a conduit. The ease and time for placement of the air-Q, fiberoptic grade of laryngeal view, time for fiberoptic tracheal intubation, and peri-operative complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA I to III) children who will be intubated as part of their general anesthesia plan for their scheduled surgeries
* Age 1 month - 2 years
* Weight 1-20 Kg

Exclusion Criteria:

* Children with active respiratory infection
* Known history of difficult mask ventilation
* Diagnosis of a congenital syndrome associated with difficult airway management
* Airway abnormalities (e.g., laryngomalacia, subglottic stenosis).

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time for successful fiberoptic tracheal intubation | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The time for successful intubation will be from removal of the face mask or disconnection of the circuit from the air-Q until evidence of end-tidal CO2 is confirmed.

SECONDARY OUTCOMES:
Time to successful placement of the Air-Q | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Successful placement of the air-Q will start with the removal of the facemask until presence of end-tidal CO2 is confirmed.
Number of attempts to place the Air-Q | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Number of attempts needed for successful placement will be recorded (maximum of 3 attempts will be considered as a failure)
Ease for placement of the air-Q | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The ease for Air-Q placement will be assessed using a subjective scale
Fiberoptic grade of laryngeal view | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The laryngeal alignment through the devices will be graded using an established scoring system
Peri-operative complications | Measured at 24 hours after device placement/study initiation
  Includes: Complications during the placement of the Air-Q (Laryngospasm, Bronchospasm, Desaturation, etc. Oropharyngolaryngeal morbidity at discharge, participants will be followed for the duration of anesthesia and after surgery, an average of 24 hours. Oropharyngolaryngeal morbidity at 24 hours post-operatively, measured at 24 hours after device placement/study initiation. These will be assessed by the subject's response or parents subjective assesment to standardized questions regarding oropharyngeal complaints such as sore throat, jaw pain, neck discomfort.
Number of attempts for fiberoptic tracheal intubation | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Number of attempts needed for successful fiberoptic tracheal intubation will be recorded (maximum of 3 attempts will be considered as a failure)
Ease for fiberoptic tracheal intubation | Participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The ease for fiberoptic tracheal intubation will be assessed using a subjective scale

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Lisa Sohn, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Hodzovic I, Janakiraman C, Sudhir G, Goodwin N, Wilkes AR, Latto IP. Fibreoptic intubation through the laryngeal mask airway: effect of operator experience*. Anaesthesia. 2009 Oct;64(10):1066-71. doi: 10.1111/j.1365-2044.2009.06030.x. PMID 19735396
- [Background] Hodzovic I, Petterson J, Wilkes AR, Latto IP. Fibreoptic intubation using three airway conduits in a manikin: the effect of operator experience. Anaesthesia. 2007 Jun;62(6):591-7. doi: 10.1111/j.1365-2044.2007.05054.x. PMID 17506738
- [Background] Erb T, Marsch SC, Hampl KF, Frei FJ. Teaching the use of fiberoptic intubation for children older than two years of age. Anesth Analg. 1997 Nov;85(5):1037-41. doi: 10.1097/00000539-199711000-00013. PMID 9356095
- [Background] Jagannathan N, Kozlowski RJ, Sohn LE, Langen KE, Roth AG, Mukherji II, Kho MF, Suresh S. A clinical evaluation of the intubating laryngeal airway as a conduit for tracheal intubation in children. Anesth Analg. 2011 Jan;112(1):176-82. doi: 10.1213/ANE.0b013e3181fe0408. Epub 2010 Nov 16. PMID 21081777